CLINICAL TRIAL: NCT01368497
Title: Clinical Trial of Entecavir/Pegylated Interferon in Immune Tolerant Children With Chronic HBV Infection (HBRN)
Brief Title: Entecavir/Pegylated Interferon in Immune Tolerant Children With Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK082864 HBRN IT Peds Trial; U01DK082916 (NIH); U01DK082864 (NIH); U01DK082874 (NIH); U01DK082944 (NIH); U01DK082843 (NIH); U01DK082871 (NIH); UL1TR000423 (NIH); UL1TR000004 (NIH); A-DK-3002-001 (Other: Interagency agreement with NIDDK)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; HBV
MeSH Terms: conditions — Hepatitis B | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entecavir and peginterferon (Experimental): Entecavir for 8 weeks followed by 40 weeks of both entecavir and peginterferon
  Interventions: Drug: Entecavir and peginterferon

INTERVENTIONS:
Drug: Entecavir and peginterferon — Entecavir 0.015 mg/kg/day (up to 0.5 mg maximum daily dose) once daily for 48 weeks and Peginterferon alfa-2a 180 µg/1.73m2 subcutaneously once weekly for 40 weeks beginning 8 weeks after entecavir monotherapy).
  Other Names: PEGASYS, peginterferon alfa 2a, Baraclude

SUMMARY:
The purpose of this study is to determine the safety and efficacy of treatment using a combination of drugs (entecavir and pegylated interferon) in children ages 3-<18 years old with immunotolerant chronic hepatitis B.

DETAILED DESCRIPTION:
This single arm treatment study was conducted by the pediatric centers within the National Institute of Diabetes Digestive and Kidney Diseases (NIDDK)-sponsored Hepatitis B Research Network (HBRN). Children age 3-<18 years with immunotolerant chronic hepatitis B (CHB) infection who fulfilled the entry criteria received entecavir as monotherapy for 8 weeks and then combination therapy with entecavir and pegylated interferon by weekly subcutaneous injection until week 48. Children were to be followed for 48 weeks after discontinuation of therapy (week 96 for those who completed 48 weeks of treatment).

Assessment was undertaken at baseline, weeks 4, 8, 10, 12, 14, & 16, then every 4 weeks until week 48, and then 4, 8, 12, 24,36, and 48 weeks following treatment discontinuation corresponding to weeks 52, 56, 60, 72, 84 and 96 for those who received treatment for 48 weeks. Blood work was drawn to measure markers of viral and liver disease status and for research biospecimen banking.

Participants were to receive therapy until week 48 and enter 48 weeks of follow-up thereafter. Participants who experienced a sustained elevation of alanine aminotransferase (ALT) were eligible to receive treatment as recommended by their hepatologist and continued to complete the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in & completed the baseline evaluation in NCT01263600 OR completed necessary components of NCT01263600 baseline evaluation by the end of the baseline visit.
* 3 to <18 years at time of randomization (day 0).
* Documented chronic Hepatitis B virus (HBV) infection as evidenced by detection of hepatitis B surface antigen (HBsAg) in serum for ≥ 24 weeks prior to baseline OR positive HBsAg and negative anti-Hepatitis B core (HBc) immunoglobulin (IgM) within 24 weeks of baseline visit.
* Presence of hepatitis B e-antigen (HBeAg) in serum at the last screening visit within 6 weeks of baseline visit.
* Serum HBV DNA level >10^7 IU/mL on at least 2 occasions at least 12 weeks apart during the 52 weeks before baseline visit. The HBV DNA levels must be within 6 weeks of baseline visit.
* ALT ≤60 U/l in males or ≤40 U/l in females, measured on at least 2 occasions, at screening (within 6 weeks prior to baseline visit) & at least 12 weeks prior to the screening visit & within the 52 weeks prior to baseline visit.
* Compensated liver disease, with normal total bilirubin (except if Gilbert's syndrome), direct bilirubin ≤0.5 mg/dL, International Normalized Ratio (INR) ≤1.5, and serum albumin ≥3.5 g/dL.
* Creatinine clearance 90 ml/min.
* Absence of hepatocellular carcinoma on liver ultrasound in the past 48 weeks.

Exclusion criteria:

* Presence of infection with Hepatitis C virus (HCV)-RNA or anti-HCV, anti-Hepatitis D virus (HDV), or HIV at screening.
* Presence of another cause of liver disease or hepatocellular cancer (HCC) (serum alpha-fetoprotein >50ng /ml).
* Evidence of decompensated liver disease (Childs B-C).
* History or other evidence of a medical condition associated with chronic liver disease (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures).
* Females who are pregnant or breastfeeding.
* Adolescent females unwilling or unable to use an acceptable method of contraception if sexually active during the treatment period.
* Children currently breastfeeding while their mother is taking lamivudine, or those who were exposed to lamivudine for ≥24 weeks via maternal lamivudine treatment during pregnancy and/or while breastfeeding.
* Previous liver or other organ transplantation including engrafted bone marrow transplant.
* Hematological abnormalities during the screening period that contraindicate full dosing with study drugs, e.g absolute neutrophil count < 1.5 x 10^9 cells/L or platelet count < 120 x 10^9 cells/L.
* Known allergy to study drugs; peginterferon alfa-2a or entecavir.
* Treatment with systemic acyclovir or famciclovir within the previous 6 months.
* Need for ongoing use of any antivirals with activity against HBV during the course of the study or history of receiving treatment for HBV.
* Any use of illegal drugs OR use of alcoholic beverages which in the opinion of a study physician is sufficient to prevent adequate compliance with study procedures or increase the risk of pancreatitis or hepatotoxicity.
* History of immunologically mediated disease (e.g. inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune haemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis).
* History or other evidence of bleeding from esophageal varices or consistent with decompensated liver disease.
* History or other evidence of chronic pulmonary disease associated with functional limitation.
* History of significant cardiovascular diseases.
* History of a severe seizure disorder or current anticonvulsant use.
* History or other evidence of severe retinopathy.
* History of thyroid disease poorly controlled on prescribed medications. Participants with elevated thyroid stimulating hormone concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease are excluded.
* Concomitant use or use during ≤ 6 months prior to the first dose of study drug of anti-neoplastic, immunosuppressive, nephrotoxic or hepatotoxic medication, methadone, theophylline or medications that may affect renal excretion or hepatic metabolism are not permitted.
* Concomitant use of complementary or alternative medications purported to have antiviral activity.
* A participant may not be co-enrolled in another clinical trial where an investigational drug is administered.
* Any other condition or situation that in the opinion of a study physician would make the participant unsuitable for enrollment or could interfere with the participant participating in and completing the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Averell Sherker, MD, Study Chair — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Ed Doo, MD, Study Chair — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Kathleen Schwarz, MD, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (6):
  - University of California San Francisco Medical Center, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis Children's Medical Center, St Louis, Missouri
  - University of Texas Southwestern, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital of Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All data will be sent to the NIDDK-supported data repository.
Supporting Information: Study Protocol, SAP
Time Frame: At completion of HBRN project. Length of availability determined by NIDDK data repository.
Access Criteria: Per NIDDK-supported data repository.

REFERENCES:
- [Background] Morris NM, Udry JR. Validation of a self-administered instrument to assess stage of adolescent development. J Youth Adolesc. 1980 Jun;9(3):271-80. doi: 10.1007/BF02088471. PMID 24318082
- See also: Click here for more information about the Hepatitis B Research Network — http://www.hepbnet.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty children were enrolled at 7 pediatric clinical sites in the United States and Canada between 9/20/2012 and 12/30/2014.
Groups:
- Entecavir and Peginterferon: Entecavir 0.015 mg/kg/day (up to 0.5 mg maximum daily dose) once daily for 48 weeks and Peginterferon alfa-2a 180 μg/1.73m^2 subcutaneously times the participant's body surface area once weekly during weeks 9-48 of treatment. After treatment discontinuation, follow-up off treatment for 48 weeks.
Period: Overall Study
Arm/Group | Entecavir and Peginterferon
Started | 60
End of Treatment | 60 (Five discontinued study drugs early and completed the follow-up period per protocol.)
Completed | 58
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 10.9 [3.4 to 17.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1
  Black/African-American | 3
  Asian | 54
  Mixed | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 12
  United States | 48
HBV DNA [Median (Full Range); unit: log10 IU/mL] | 8.2 [7.5 to 9.1]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Hepatitis B e Antigen (HBeAg) Loss & Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Levels ≤1,000 International Units (IU) Per Milliliter (mL)
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

2. Primary Outcome: Incidence of Adverse Events (AEs) Per Person-Year
Description: The number of AEs includes both AEs and Serious Adverse Events (SAEs). The incidence is calculated as the number of AEs divided by the number of person-years of observation, which is the sum, across all participants, of the number of years between the start of treatment and the end of treatment, or the end of follow-up, respectively.
Time Frame: From first treatment to the end of treatment (up to 48 weeks) and the end of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: AEs per person-year of observation
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
AEs per person-year of observation
  End of treatment (Up to 48 weeks) | 1.13 [0.88 to 1.46]
  End of follow-up (Up to 96 weeks) | 0.70 [0.56 to 0.87]

3. Primary Outcome: Incidence of Serious Adverse Events (SAEs) Per Person-Year
Description: The incidence is calculated as the number of SAEs divided by the number of person-years of observation, which is the sum, across all participants, of the number of years between the start of treatment and the end of treatment, or the end of follow-up, respectively.
Time Frame: From first treatment to the end of treatment (up to 48 weeks) and the end of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: SAEs per person-year of observation
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
SAEs per person-year of observation
  End of treatment (Up to 48 weeks) | 0 [NA to NA] — 95% Confidence Interval (CI) around 0 not calculated
  End of follow-up (Up to 96 weeks) | 0.01 [0.00 to 0.07]

4. Secondary Outcome: Proportion of Participants With Hepatitis B Surface Antigen (HBsAg) Loss
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .050 [.010 to .139]

5. Secondary Outcome: Proportion of Participants With Hepatitis B Surface Antigen (HBsAg) Loss
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

6. Secondary Outcome: Proportion of Participants With Hepatitis B e Antigen (HBeAg) Loss
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

7. Secondary Outcome: Proportion of Participants With Hepatitis B e Antigen (HBeAg) Loss
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

8. Secondary Outcome: Proportion of Participants With HBeAg Seroconversion
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

9. Secondary Outcome: Proportion of Participants With HBeAg Seroconversion
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

10. Secondary Outcome: Proportion of Participants With HBsAg Seroconversion
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

11. Secondary Outcome: Proportion of Participants With HBsAg Seroconversion
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

12. Secondary Outcome: Proportion of Participants With Alanine Aminotransferase (ALT) ≤ 40 Units (U) Per Liter (L) for Males, ≤ 35 U/L for Females
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .350 [.231 to .484]

13. Secondary Outcome: Proportion of Participants With ALT ≤ 40 U/L for Males, ≤ 35 U/L for Females
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .650 [.516 to .769]

14. Secondary Outcome: Proportion of Participants With HBV DNA ≤1000 IU/mL
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .750 [.621 to .853]

15. Secondary Outcome: Proportion of Participants With HBV DNA ≤1000 IU/mL
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

16. Secondary Outcome: Proportion of Participants With HBV DNA < 20 IU/mL
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .233 [.134 to .360]

17. Secondary Outcome: Proportion of Participants With HBV DNA < 20 IU/mL
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .033 [.004 to .115]

18. Secondary Outcome: Proportion Without Detectable Antiviral Drug-resistance HBV Mutations
Description: HBV drug resistance variant testing was performed at the CDC laboratory. The sequences of the HBV polymerase spanning nucleotide positions 311-1021 were determined by Sanger sequencing. Drug resistance mutations that were tested in this study included L80VI, L82M, T128N, W153Q, F166L, I169T, V173L, L180M, A181TV, T184ACFGILMS, V191T, A194T, A200V, S202ETV, M204IV, V207I, N236T, M250ILV, and G145R.
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Proportion of participants | .733 [.603 to .839]

19. Secondary Outcome: Growth Measures: Z-scores Weight, Height, and Body Mass Index
Description: A child's Z-score is the number of standard deviations that the child is from the average of children of the same sex and age from a reference population. The reference population is provided in the 2000 Centers for Disease Control and Prevention (CDC) growth charts. Positive Z scores mean the growth measure (weight, height, or body mass index) is above the average, negative Z scores mean the growth measure is below the average.
Time Frame: End of treatment (up to 48 weeks)
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Z-score
  Z-score weight | -0.48 [-0.94 to -0.10]
  Z-score height | -0.41 [-0.78 to -0.04]
  Z-score BMI | -0.37 [-0.82 to 0.01]

20. Secondary Outcome: Growth Measures: Z-scores Weight, Height, and Body Mass Index
Description: as for outcome 19
Time Frame: End of follow-up (up to 96 weeks)
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Z-score
  Z-score weight | -0.34 [-0.81 to 0.02]
  Z-score height | -0.45 [-0.88 to -0.04]
  Z-score BMI | -0.14 [-0.54 to 0.21]

21. Secondary Outcome: Tanner Stages of Physical Growth
Description: The Tanner Stage questionnaire is only completed by participants 8 years of age and older. The copyrighted form includes pictures and descriptions. Girls selected the picture closest to their self-perceived breast growth from among 5 stages of breast growth and boys did the same for testes, scrotum, and penis growth.
  Boys: I-prepubertal; II-enlargement of scrotum and testes; III-enlargement of the penis and further growth of testes; IV- increased size of penis with growth in breadth and development of glans, testes, and scrotum larger, scrotum skin darker; V- adult genitalia.
  Girls: I-prepubertal; II-breast bud stage with the elevation of breast and papilla and enlargement of the areola; III-further enlargement of breast and areola, no separation of their contour; IV-areola and papilla form a secondary mound above the level of the breast; V: mature adult stage.
  There is no "better" or "worse" outcome. They are self-assessed descriptive measures of physical growth.
Time Frame: End of treatment (up to 48 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Participants
  I | 12
  II | 3
  III | 12
  IV | 8
  V | 7
  Missing | 18

22. Secondary Outcome: Tanner Stages of Physical Growth
Description: as for outcome 21
Time Frame: End of follow-up (up to 96 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Participants
  I | 14
  II | 5
  III | 9
  IV | 8
  V | 12
  Missing | 12

23. Secondary Outcome: Tanner Stages of Pubic Hair Growth
Description: The Tanner Stage questionnaire is only completed by participants 8 years of age and older. The copyrighted form includes pictures and descriptions. Participants selected the picture closest to their self-perceived pubic hair growth.
  Boys and girls: I-prepubertal (no pubic hair at all); II-sparse growth of long, slightly pigmented hair, straight or curled, at base of penis or along labia; III: darker, coarser and more curled hair, spreading sparsely over junction of pubes; IV- hair adult in type, but covering smaller area than in adult; V-adult in type and quantity.
  There is no "better" or "worse" outcome. They are self-assessed descriptive measures of physical growth.
Time Frame: End of treatment (up to 48 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Participants
  I | 15
  II | 4
  III | 4
  IV | 12
  V | 7
  Missing | 18

24. Secondary Outcome: Tanner Stages of Pubic Hair Growth
Description: as for outcome 23
Time Frame: End of follow-up (up to 96 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Entecavir and Peginterferon
Number analyzed (Participants) | 60
Participants
  I | 16
  II | 6
  III | 5
  IV | 9
  V | 12
  Missing | 12

ADVERSE EVENTS:
Time Frame: Study entry (consent) to the end of follow-up (48 weeks following the end of treatment).
Description: Expected symptoms/signs or common side effects of study meds need not be reported (these are Adverse Effects). These are a guide for recording adverse events, which are at the discretion of the investigator.
  1. Symptom or event requiring discontinuation of study medication.
  2. New symptom or event requiring a written prescription for treatment.
  3. New symptom or event resulting in a referral to another provider.
  4. Grade 3 or 4 event per the NCI Common Toxicity Criteria.
Arm/Group | Entecavir and Peginterferon
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 37/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entecavir and Peginterferon (N=60)
Myasthenia gravis (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entecavir and Peginterferon (N=60)
Small splenic mass (Blood and lymphatic system disorders) | 1 (1)
Low absolute neutrophil count (Blood and lymphatic system disorders) | 10 (13)
Low absolute neutrophil count and platelets (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Syncope Episode (Cardiac disorders) | 1 (1)
Fluid in left ear (Ear and labyrinth disorders) | 1 (1)
Thyroid-stimulating hormone (TSH) elevation (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Bilateral conjunctivitis (Eye disorders) | 1 (1)
Blurry vision (Eye disorders) | 1 (1)
Decreased visual acuity (Eye disorders) | 1 (2)
Upset stomach (Gastrointestinal disorders) | 1 (1)
Elective extraction of four primary teeth (General disorders) | 1 (1)
Nauseous and achy (General disorders) | 1 (1)
Mild nose bleed (General disorders) | 1 (2)
Sore throat (General disorders) | 1 (1)
ALT or AST elevation (Hepatobiliary disorders) | 6 (6)
Total bilirubin elevation (Hepatobiliary disorders) | 1 (2)
Bilateral periocular dermatitis (Immune system disorders) | 1 (1)
Bilateral rash and swelling of feet (Immune system disorders) | 1 (1)
Hives (Immune system disorders) | 1 (1)
Strep throat (Infections and infestations) | 4 (4)
Ear infection (Infections and infestations) | 1 (1)
Infection from tooth extraction (Infections and infestations) | 1 (1)
Keratitis and uveitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinus infection (Infections and infestations) | 4 (5)
Sore throat and fever (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Creatinine elevation (Metabolism and nutrition disorders) | 1 (1)
Creatine kinase elevation (Musculoskeletal and connective tissue disorders) | 1 (1)
Ptosis (Nervous system disorders) | 1 (1)
Febrile seizure (Nervous system disorders) | 1 (1)
Short temper or slight agitation (Psychiatric disorders) | 1 (2)
Occult blood in urine (Renal and urinary disorders) | 1 (1)
Menstrual cramping (Reproductive system and breast disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Abscess gum from tooth extraction (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
From the Publications and Presentations policy "Disagreements between the HBRN Steering Committee and the NIDDK on the merits of journal submission of a specific manuscript will be mediated through discussion on Steering Committee conference calls, ad hoc conference calls or during face to face Steering Committee meetings. The decision of the NIDDK is final and cannot be appealed."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT01368497/Prot_SAP_000.pdf